CLINICAL TRIAL: NCT05555160
Title: Application of Intracavity Electrocardiogram Positioning Technique in Catheterization of Valvular PICC
Brief Title: Application of Intracavity Electrocardiogram Positioning Technique in PICC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong Branden Med.Device Co.,Ltd (Industry)
Collaborators: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-202103
Record Dates: First submitted 2021-09-22; First posted 2022-09-26 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2021-09

CONDITIONS: Patients Requiring Peripherally Inserted Central Venous Catheters

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-chamber valve tip conductive PICC catheter (Experimental)
  Interventions: Device: PICC
- Single - chamber valve non - tip conductive PICC catheter (Experimental)
  Interventions: Device: PICC

INTERVENTIONS:
Device: PICC — Peripheral central venous catheterization (PICC) is mainly applied to patients with medium and long-term intravenous infusion, infusion of stimulant drugs and intermittent infusion of chemotherapy drugs. It is a catheterization technology to place PICC through peripheral veins and make its tip reach the central vein

SUMMARY:
This study was a prospective, multicenter, randomized controlled study. The study aimed to exploring the influence of PICC intra catheter guide wire or PICC conductive tip as intra luminal electrode on the positioning accuracy of catheter tip and exploring the influence of PICC intra catheter guide wire or PICC conductive tip as intra luminal electrode on catheterization complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old who need PICC catheterization for the first time according to the doctor's advice;
* No serious cardiovascular diseases before catheterization, such as atrial fibrillation, pulmonary heart disease and other P wave abnormalities, serious heart block, etc.;
* patients who did not participate in other clinical studies;
* Patients who voluntarily participated in the clinical study, signed informed consent and cooperated with clinical follow-up

Exclusion Criteria:

* patients with local malformation or scar formation;
* Patients with infection or damage at the puncture site;
* patients with tumor compression of blood vessels;
* Patients with confirmed or suspected catheter-related infection, bacteremia and septicemia
* Patients diagnosed or suspected to be allergic to silicone material
* Patients with a history of radiotherapy at the pre-intubation site
* Patients with a history of venous thrombosis, trauma or vascular surgery
* Patients with superior vena cava syndrome
* Patients with poor medical behavior
* Patients with severe peripheral vascular edema
* High-flow fluid infusion, patients requiring hemodialysis, pacemaker installation, crutches, or patients who may undergo A-V fistula

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3051 (Estimated)
Dates: Start 2022-09-30 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of tip determination | Immediately after surgery
  IC-ECG method was used to place the tube, and X-ray was used to determine the accuracy of tip location after confirmation. If the two judgments are inconsistent, the third method, such as echocardiography, shall be used. The tip determination accuracy of IC-ECG localization method and X-ray localization method were calculated respectively.X-ray judgment standard: the reference standard is the first choice of the cardiac shadow method: not exceeding the highest protrusion on the left side of the cardiac shadow (tracheal protrusion method: 0-3cm below the tracheal protrusion); Secondary rib reading method: posterior 5-7 ribs.

SECONDARY OUTCOMES:
incidence of PICC-related complications | After the operation to 180 days
  Complications related to puncture and catheter during tube placement and retention include redness and swelling, bleeding, exudation, puncture point infection, ectopic catheter, displacement, catheter blockage, rupture, phlebitis and thrombosis.
success rate of one catheterization | Immediately after surgery
  one-time successful catheterization means that the tip of the catheter can be placed at the ideal position in one catheterization operation, without adjustment after X-ray confirmation. After catheterization, both groups of patients need to verify whether the tip is in the ideal position through X-ray, and whether the operation is successful also needs to be judged through X-ray, and the X-ray results need to be retained (random number, center code, initials, time). All results will be sent to the central laboratory for analysis and interpretation.
rate of convenient | Immediately after surgery
  survey whether the operators think the operation is convenient through questionnaires made by ourselves.
rate of unplanned extubation | After the operation to 180 days
  Proportion of early removal due to complications
Retention duration | After the operation to 180 days
Medical costs resulting from complications | After the operation to 180 days

IPD SHARING:
Plan to Share IPD: Undecided